CLINICAL TRIAL: NCT05578066
Title: Reducing Stigma Toward Mental Illness and Substance Use Issues in Primary Health Care in Chile: A Cluster Randomized Control Trial.
Brief Title: Reducing Stigma Toward Mental Illness and Substance Use Issues in Primary Health Care in Chile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FONDECYT 1201504
Record Dates: First submitted 2022-05-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-05

CONDITIONS: Mental Health; Substance Abuse; Stigmatization
Keywords: Primary Health Care; Implementation science; social stigma
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Stereotyping; Social Stigma

STUDY DESIGN:
Intervention Model Description: A two-arm, cluster-randomized controlled trial with CESFAMs being the unit of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will be composed by aproximately 8 CESFAM with 36 Primary Health Care providers that are currently employed with a total of 288 providers per arm. And some PHC users that have received care there for Mental Health Abuse Issues in the three months prior to study participation.
  The interventions include a comprehensive, 18-month, recovery-oriented anti-stigma intervention is composed by five components.
  1. Developing a Team of Local Champions
  2. Analysis of Internal Policies, Procedures and Protocols
  3. Raising Awareness
  4. Innovative Contact-Based Education
  5. Recovery based Arts.
  Teams of leaders developed as part of the first component will assist the research team with the implementation of the anti-stigma intervention at their respective CESFAM.
  Interventions: Other: Developing teams of Local Leaders; Other: Analysis of Internal Policies, Procedures and Protocols; Other: Raising Awareness; Other: Innovative Contact-Based Education; Other: Recovery-Based Arts
- Control group (No Intervention): The control group will be composed by aproximately 8 CESFAM with 36 Primary Health Care providers that are currently employed with a total of 288 providers per arm. And some PHC users that have received care there for Mental Health Abuse Issues in the three months prior to study participation.
  Data will be collected from this group in order to generate an integrated analysis with the information recolected from the intervention group.

INTERVENTIONS:
Other: Developing teams of Local Leaders — A team of local leaders, consisting of 3-5 PHC providers and 1-2 users at each CESFAM will be developed in months 1-3 of the intervention.The teams will comprise some individuals who have provided critical support and input, including participating in the exploratory research phase and the Community-Based Participatory Research (CBPR) adaptation of the intervention framework for the Chilean context developed previously. The teams will assist with the data collection process throughout the study by encouraging colleagues to complete questionnaires and recruit users, as well as oversee and implement the intervention at their respective CESFAM. They will receive training to develop their skills as leaders and support the implementation process at their respective CESFAM.
  Arms: Intervention group
Other: Analysis of Internal Policies, Procedures and Protocols — This component involves evaluating CESFAM policies, procedures, and protocols using an anti-stigma/pro-recovery approach to identify strengths and areas for improvement in service delivery for individuals affected by MISUI. This will be completed using a policy analysis tool based on existing frameworks, such as the Health Equity Impact Assessment Tool (PHO & OMHLTC, 2012) and the QualityRights Toolkit (WHO, 2012). At least 5 policies, procedures, or protocols to be analyzed will be selected by the local leaders at intervention CESFAM during months 3-6 of the intervention. Recommendations concerning health equity, prevention of stigma, and promotion of recoveryoriented practices for individuals with MISUI will be developed and shared following analysis. Each intervention CESFAM will be expected to implement at least one recommendation and make the necessary efforts to educate PHC providers about the policy change in months 7-18 of the intervention.
  Arms: Intervention group
Other: Raising Awareness — Various forms of media will be used to raise awareness about stigma related to MISUI among PHC providers and users. Local leaders at intervention CESFAM will determine the type of media they would like to use; this may include images, film, music, or a combination of media. The research team will work with local leaders to develop messaging to include in the media and assist with showcasing these pieces within each intervention CESFAM. This component will be implemented throughout the intervention (intervention months 1-18). Depending on the type of media, instances of use will be tracked accordingly. For example with posters, data on the number of posters posted at a CESFAM over what time period and an estimation of the number of PHC providers and users who have viewed the posters will be collected.
  Arms: Intervention group
Other: Innovative Contact-Based Education — Educational workshops will include anti-stigma and recovery principles, along with specific MISUI topics relevant to PHC providers. This will be determined by findings from the exploratory phase, current research, best practices, and the perspectives of local leaders. It may include (1) supporting CESFAM PHC providers in preventing stigma and promoting recovery in their practice and (2) enhancing the competencies of CESFAM PHC providers for discussing MISUI with their users, identifying MISUI signs and symptoms, and referring users to psychosocial centres for treatment. The key feature of these workshops is the contact-based educational element, where people with lived experience participate in developing and delivering the curriculum to CESFAM PHC providers. Four three-hour workshops will be held at each intervention CESFAM and will be facilitated by two academic/clinical trainers with expertise in stigma research and practice, and one person with lived experience.
  Arms: Intervention group
Other: Recovery-Based Arts — Local leaders at CESFAM will select one PHC provider member and recruit one artist to develop an arts curriculum and facilitate the art sessions. The facilitators will select an art form to use throughout the sessions, and in collaboration with local leaders they will determine themes related to MISUI to cover in each session (planning process will be completed in intervention months 7-8). Arts workshops will be held for 10 weeks, with each session lasting up to three hours (during intervention months 9-12). Ten users affected by MISUI and at least three CESFAM PHC providers will participate in the workshops each week. At the end of the 10-week program, each CESFAM will host an exhibition to showcase the artwork that has been produced (during intervention months 13-18). All PHC providers and users, as well as community members, will be invited to attend the exhibition. PHC providers and users will be invited to speak about their experiences learning and working together to create art.
  Arms: Intervention group

SUMMARY:
This research project aims to determine the effectiveness of a comprehensive anti-stigma intervention in reducing stigmatizing attitudes and behaviours among Primary Health Care (PHC) providers toward individuals with mental illness and/or substance use issues (MISUI) in the Chilean context, using Centros de de Salud Familiar (CESFAMs) as the point of intervention.

DETAILED DESCRIPTION:
The intervention model will be culturally adapted with CESFAM PHC provider and user input to be relevant and valid to Chile. The 18-month intervention includes five (5) components that are simultaneously implemented in CESFAMs: (1) Develop a Team of Local Champions in each intervention CESFAM, comprising PHC providers and users; (2) Analysis of Internal CESFAM Policies, Procedures, and Protocols to determine areas of improvement in service delivery for individuals with MISUI; (3) Raising Awareness of stigma toward MISUI using various forms of media within the CESFAM; (4) Innovative Contact-Based Education workshops on anti-stigma and recovery principles, co-lead by academic/clinical trainers and a person with lived experience of MISUI; and (5) Recovery-Based Arts, a multi-week arts workshop for PHC providers and users to produce artwork related to MISUI and recovery, culminating in an exhibition to showcase artwork for the CESFAM providers, users, and community.

Due to Coronavirus disease of 2019 (COVID-19) sanitary context some of the interventions may be developed remotly dependind on each primary healthcare center needs and capability. This interventions will be implemented in years two and three of the study and the final year of the study is dedicated to integrated data analysis, a 6-month follow-up data collection, and dissemination of results.

If the intervention proves to be effective, control CESFAMs will be provided with an anti-stigma initial training and protocols for intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* CESFAM must serve a registered population of at least 15,000 people
* CESFAM have at least 50 staff employed

Exclusion Criteria:

* CESFAM being part of another antistigma program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Survey for PHC Providers (Scale 1 - main scale) | 2 years
  A self-administered questionnaire will be used to examine stigma directed at persons with MISUI among health professionals. This questionnaire will be completed at four time-points (baseline, mid-point, end-point, and 6-month follow-up). It will collect data related to two main components: (1) socio-demographic and other relevant general variables (see Appendix 1.10 for variables); and (2) attitudes toward MISUI stigma and recovery. The end-point questionnaire will also include a third component focusing on the intervention and its implementation.
  The main scale to measure stigma toward MISUI to include in the questionnaire is the Opening Minds Scale for Health Care Providers (OMS-HC6). This 20-item instrument can result in a possible score of 20 to 100, with a higher score indicating more stigmatizing attitudes and behavioral intentions. Some items in the scale require reverse coding. There is also a 15-item version.
  In addition, complementing, four other scales are considered.
Survey for PHC Providers (Scale 2) | 2 years
  Mental Illness: Clinicians' Attitudes (MICA 7; overall scores range from a minimum of 16 to a maximum of 96, with higher scores indicating more stigmatizing and negative attitudes toward mental illness).
Survey for PHC Providers (Scale 3) | 2 years
  Modified Bogardus Social Distance Scale (scores from 9 to 36, higher scores represent greater social distance) or Grandon Social Distance Scale (scores from 5 to 25, higher scores represent less social distance)
Survey for PHC Providers (Scale 4) | 2 years
  Recovery Assessment Scale for Providers (Score range: 13 -least negative attitudes toward recovery- to 117 -most negative attitudes regarding recovery-).
Survey for PHC Users | 2 years
  A face-to-face survey assisted by a research team member be used to examine how users perceive stigmatizing attitudes and behaviours among CESFAM PHC providers. The questionnaire will include four main components: (1) socio-demographic and other relevant general variables; (2) perceived stigmatizing attitudes and behaviours among CESFAM PHC providers; (3) perceived recovery-oriented practices by CESFAM PHC providers; and (4) accessing healthcare at their CESFAM. The questionnaire will take approximately 30 minutes to complete. The Perceived Devaluation-Discrimination Scale will be used to assess the extent to which users believe that other people devalue or discriminate against someone with MISUI. And adapted version of the Discrimination Experience Subscale of the 29-item Internalized Stigma of Mental Illness (ISMI).
Identify critical barriers and opportunities for its implementation in PHC | 2 years
  To evaluate implementation of the intervention, qualitative interviews will be held with two PHC providers (local champions) and one CESFAM authority per intervention site at baseline, mid-point, and end-point. In addition, at least one local champion from the community will be interviewed to explore his/her experience as a leader, pros and cons of the intervention and how it could be improved. Questions will relate to implementation outcomes for the intervention: acceptability, adoption, appropriateness, feasibility, fidelity, implementation cost, coverage and sustainability.
  The Consolidated Framework for Implementation Research (CFIR) will be considered to guide the process.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime C Sapag, Phd, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Cesfam Chuchunco, Santiago, Chile

REFERENCES:
- [Background] Parra Videla C, Sapag JC, Klabunde R, Velasco PR, Anriquez S, Aracena Alvarez M, Mascayano F, Bravo P, Sena BF, Jofre Escalona A, Bobbili SJ, Corrigan PW, Bustamante I, Poblete F, Alvarado R. Cross-cultural adaptation of four instruments to measure stigma towards people with mental illness and substance use problems among primary care professionals in Chile. Transcult Psychiatry. 2023 Apr;60(2):286-301. doi: 10.1177/13634615221100377. Epub 2022 Jul 12. PMID 35821607
- [Background] Kassam A, Papish A, Modgill G, Patten S. The development and psychometric properties of a new scale to measure mental illness related stigma by health care providers: the Opening Minds Scale for Health Care Providers (OMS-HC). BMC Psychiatry. 2012 Jun 13;12:62. doi: 10.1186/1471-244X-12-62. PMID 22694771
- [Background] Khenti A, Mann R, Sapag JC, Bobbili SJ, Lentinello EK, Maas MV, Agic B, Hamilton H, Stuart H, Patten S, Sanches M, Corrigan P. Protocol: a cluster randomised control trial study exploring stigmatisation and recovery-based perspectives regarding mental illness and substance use problems among primary healthcare providers across Toronto, Ontario. BMJ Open. 2017 Nov 20;7(11):e017044. doi: 10.1136/bmjopen-2017-017044. PMID 29162572
- [Background] Murney MA, Sapag JC, Bobbili SJ, Khenti A. Stigma and discrimination related to mental health and substance use issues in primary health care in Toronto, Canada: a qualitative study. Int J Qual Stud Health Well-being. 2020 Dec;15(1):1744926. doi: 10.1080/17482631.2020.1744926. PMID 32228393
- [Background] Khenti A, Bobbili SJ, Sapag JC. Evaluation of a Pilot Intervention to Reduce Mental Health and Addiction Stigma in Primary Care Settings. J Community Health. 2019 Dec;44(6):1204-1213. doi: 10.1007/s10900-019-00706-w. PMID 31317439
- [Background] Khenti A, Thomas FC, Mohamoud S, Diaz P, Vaccarino O, Dunbar K, Sapag JC. Mental health and addictions capacity building for community health centres in Ontario. Can Fam Physician. 2017 Oct;63(10):e416-e424. PMID 29025818
- [Background] Sapag JC, Sena BF, Bustamante IV, Bobbili SJ, Velasco PR, Mascayano F, Alvarado R, Khenti A. Stigma towards mental illness and substance use issues in primary health care: Challenges and opportunities for Latin America. Glob Public Health. 2018 Oct;13(10):1468-1480. doi: 10.1080/17441692.2017.1356347. Epub 2017 Aug 2. PMID 28766377
- [Background] van der Maas M, Stuart H, Patten SB, Lentinello EK, Bobbili SJ, Mann RE, Hamilton HA, Sapag JC, Corrigan P, Khenti A. Examining the Application of the Opening Minds Survey in the Community Health Centre Setting. Can J Psychiatry. 2018 Jan;63(1):30-36. doi: 10.1177/0706743717719079. Epub 2017 Jun 30. PMID 28665144
- [Background] Mascayano F, Toso-Salman J, Ho YCS, Dev S, Tapia T, Thornicroft G, Cabassa LJ, Khenti A, Sapag J, Bobbili SJ, Alvarado R, Yang LH, Susser E. Including culture in programs to reduce stigma toward people with mental disorders in low- and middle-income countries. Transcult Psychiatry. 2020 Feb;57(1):140-160. doi: 10.1177/1363461519890964. Epub 2019 Dec 19. PMID 31856688
- [Background] Sapag JC, Velasco PR. [Stigma toward mental disorders and addictions: Study in Chilean primary care]. Aten Primaria. 2020 May;52(5):361-363. doi: 10.1016/j.aprim.2019.07.014. Epub 2019 Dec 9. No abstract available. Spanish. PMID 31831205
- [Background] Sapag JC, Klabunde R, Villarroel L, Velasco PR, Alvarez C, Parra C, Bobbili SJ, Mascayano F, Bustamante I, Alvarado R, Corrigan P. Validation of the Opening Minds Scale and patterns of stigma in Chilean primary health care. PLoS One. 2019 Sep 5;14(9):e0221825. doi: 10.1371/journal.pone.0221825. eCollection 2019. PMID 31487333
- [Background] Kemp CG, Jarrett BA, Kwon CS, Song L, Jette N, Sapag JC, Bass J, Murray L, Rao D, Baral S. Implementation science and stigma reduction interventions in low- and middle-income countries: a systematic review. BMC Med. 2019 Feb 15;17(1):6. doi: 10.1186/s12916-018-1237-x. PMID 30764820
- [Background] Nyblade L, Stockton MA, Giger K, Bond V, Ekstrand ML, Lean RM, Mitchell EMH, Nelson RE, Sapag JC, Siraprapasiri T, Turan J, Wouters E. Stigma in health facilities: why it matters and how we can change it. BMC Med. 2019 Feb 15;17(1):25. doi: 10.1186/s12916-019-1256-2. PMID 30764806
- [Background] Corrigan P, Schomerus G, Shuman V, Kraus D, Perlick D, Harnish A, Kulesza M, Kane-Willis K, Qin S, Smelson D. Developing a research agenda for understanding the stigma of addictions Part I: Lessons from the Mental Health Stigma Literature. Am J Addict. 2017 Jan;26(1):59-66. doi: 10.1111/ajad.12458. Epub 2016 Oct 25. PMID 27779803
- [Background] Corrigan PW, Schomerus G, Shuman V, Kraus D, Perlick D, Harnish A, Kulesza M, Kane-Willis K, Qin S, Smelson D. Developing a research agenda for reducing the stigma of addictions, part II: Lessons from the mental health stigma literature. Am J Addict. 2017 Jan;26(1):67-74. doi: 10.1111/ajad.12436. Epub 2016 Nov 22. PMID 27875626
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Gabbidon J, Clement S, van Nieuwenhuizen A, Kassam A, Brohan E, Norman I, Thornicroft G. Mental Illness: Clinicians' Attitudes (MICA) scale-psychometric properties of a version for healthcare students and professionals. Psychiatry Res. 2013 Mar 30;206(1):81-7. doi: 10.1016/j.psychres.2012.09.028. Epub 2012 Oct 16. PMID 23084597
- [Background] Grandon P, Saldivia S, Vaccari P, Ramirez-Vielma R, Victoriano V, Zambrano C, Ortiz C, Cova F. An Integrative Program to Reduce Stigma in Primary Healthcare Workers Toward People With Diagnosis of Severe Mental Disorders: A Protocol for a Randomized Controlled Trial. Front Psychiatry. 2019 Mar 7;10:110. doi: 10.3389/fpsyt.2019.00110. eCollection 2019. PMID 30899230
- [Background] Kates N, Arroll B, Currie E, Hanlon C, Gask L, Klasen H, Meadows G, Rukundo G, Sunderji N, Ruud T, Williams M. Improving collaboration between primary care and mental health services. World J Biol Psychiatry. 2019 Dec;20(10):748-765. doi: 10.1080/15622975.2018.1471218. Epub 2018 Jun 20. PMID 29722600
- [Background] Pescosolido BA, Martin JK. The Stigma Complex. Annu Rev Sociol. 2015 Aug;41:87-116. doi: 10.1146/annurev-soc-071312-145702. Epub 2015 May 4. PMID 26855471
- [Background] Moberg J, Kramer M. A brief history of the cluster randomised trial design. J R Soc Med. 2015 May;108(5):192-8. doi: 10.1177/0141076815582303. No abstract available. PMID 26022551
- [Derived] Sapag JC, Traub C, Velasco PR, Arratia T, Alvarado R, Aracena M, Poblete FC, Villarroel L, Bravo P, Alvarez-Huenchulaf C, Jofre Escalona A, Vargas-Malebran N, Bobbili S, Bustamante I, Khenti A, Corrigan PW. Reducing stigma toward mental illness and substance use issues in primary health care in Chile: Protocol of a cluster controlled trial study. Front Psychiatry. 2022 Dec 20;13:1083042. doi: 10.3389/fpsyt.2022.1083042. eCollection 2022. PMID 36606131